CLINICAL TRIAL: NCT00935454
Title: Intracorporeal Autologous Hepatocyte Matrix Implant: A New Tissue Engineering Procedure for Treatment of Hepatic Disease.
Brief Title: Hepatocyte Matrix Implant Study
Acronym: HMI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baermed (Other)
Responsible Party: Hans U. Baer, MD, Professor in Universitas Tarumanagara, Baermed Center For Abdominal Surgery
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baermed-001
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2009-07

CONDITIONS: Liver Disease; Liver Cirrhosis
Keywords: hepatocyte matrix implantation; endstage liver disease; liver cirrhosis; impaired liver parenchyma; improvement of liver function
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Hepatocyte matrix implantation — First operation:
  Removal of liver tissue and biopsy of pancreas
  Second operation:
  Implantation of hepatocyte matrix implant into small bowel mesentery
  Other Names: biocell liver; hepatocyte implant

SUMMARY:
This clinical investigation of the hepatocyte matrix implant is an evaluation blinded non-randomized and monocentric pilot study of Phase I, which is conducted as a therapeutic investigation. Randomization is not possible due to ethical and practical reasons. Pending approval of the ethical committee the study will also be conducted in Indonesia.

This new treatment procedure has already been successfully used on the basis of compassionate use in Germany. The hepatocyte matrix implant is a new patented procedure consisting of bio-matrix technology. A formaldehyde-free special matrix consisting of self-dissolving polymers is applied as a carrier substance and is cultivated with human autologous cells using a special technique. Clinically the bioartificial liver replacement tissue for patients with end-stage hepatic disease has been developed as a first application. In this procedure autologous hepatocytic tissue and pancreatic tissue is removed (liver resection and pancreatic biopsy) from the patient in a first surgical procedure. The tissue is sent to a specialized Cell Culture Laboratory. The laboratory is GMP certified for this procedure. The cells are processed according to SOPs in a special perfusion procedure and prepared on several platelets of matrices (platelets of 20 mm diameter and 4mm thickness). After completion of the laboratory process the biotissues are implanted into the mesentery of the small intestine during a second operation. The cells are growing controlled on the matrix, take on the capillaries of the patient and thus connect to the blood circulation. The implanted cells multiply by a specific factor and independently take over the metabolic function of the original liver after two to four weeks. In the following process the carrier matrix dissolves completely and implanted cells develop into liver cell tissue.

ELIGIBILITY:
Main Inclusion Criteria:

* endstage liver disease
* stable and non-improving liver condition for at least 3 month
* alcoholic liver cirrhosis: proven alcohol abstinence for 6 month or more
* patient in bad general condition

Main Exclusion Criteria:

* pregnancy
* drug addiction (except alcohol)
* psychiatric disease
* HIV positive
* sepsis
* peritoneal carcinosis
* hereditary liver disease
* acute liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-09 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Liver function Postoperative complication | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Baermed Center For Abdominal Surgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- See also: Center For Abdominal Surgery, Hirslanden Hospital — http://www.baermed.ch